CLINICAL TRIAL: NCT04695470
Title: Phase II Trial of Fruquintinib With Sintilimab in Treating Refractory Metastatic Colorectal Cancer Patients With TMB(Tumor Mutation Burden)-High and Non-MSI(Microsatellite Instability)-High
Brief Title: Phase II Trial of Fruquintinib With Sintilimab in Treating Selected Refractory Metastatic Colorectal Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aiping Zhou (Unknown)
Responsible Party: Sponsor-Investigator, Aiping Zhou, Professor Department of Medical Oncology Cancer Institute & Hospital Chinese Academy of Medical sciences & Peking Union Medical College (CAMS & PUMC), Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2091
Record Dates: First submitted 2021-01-04; First posted 2021-01-05 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HMPL-013; sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fruquintinib with Sintilimab (Experimental): Patients who met the eligibility criteria took fruquintinib 5mg qd for 2 weeks on and 1 week off Q3w plus Sintilimab 200mg iv, Q3w.
  Interventions: Drug: Fruquintinib and Sintilimab

INTERVENTIONS:
Drug: Fruquintinib and Sintilimab — fruquintinib 5mg qd for 2 weeks on and 1 week off, Q3w
  Sintilimab 200mg iv, Q3w

SUMMARY:
This is a prospective, Single arm Phase II trial. Patients were eligible to participate when they had histological or cytological confirmed metastatic colorectal adenocarcinoma Non-MSI(microsatellite instability)-high and TMB(tumor mutational burden)-High.

Patients had to have received at least a second-line standard therapy, including fluoropyrimidine, oxaliplatin, or irinotecan-based regimens and VEGF(vascular endothelial growth factor) inhibitors and to have disease progression within 3 months after the last administration of the last standard therapy or to have stopped such therapy due to unacceptable toxicities. Pre-treatment with anti-EGFR(epidermal growth factor receptor) were mandatory if RAS(Rat sarcoma virus) wild and left side .

Patients who met the eligibility criteria took fruquintinib plus Sintilimab until disease progression, death, unacceptable toxicity, withdrawal of consent by the patient, or decision by the treating physician that discontinuation would be in the patient's best interest. The primary study endpoint was PFS(progression free survival) rate at 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the study and signed the Informed Consent Form (ICF) out of their own will;
2. Histologically or cytologically diagnosed with metastasis colorectal adenocarcinoma CRC (Phase IV)
3. MSS or MSI-low, MSI was assessed per local guidelines (immunohistochemistry and/or polymerase chain reaction [PCR]) prior to screening. Tumor samples with instability in 0 or 1 marker were identified as microsatellite-stable and MSI-low, respectively.
4. TMB≥5 mutations/Mb, TMB was performed on plasma samples by NGS.
5. Subjects who failed at least second line standard chemotherapies including Fluorouracil, Oxaliplatin, Irinotecan and VEGF inhibitors(e.g., bevacizumab). Pre-treatment with anti-EGFR(e.g., cetuximab) were mandatory if RAS wild and left side. Failed therapies are defined as the occurance of PD or intolerable toxicities during the treatment or within 3 months after the last dose.
6. Subject must not receive any systematically anti-tumor therapies during the last 4 weeks, and never receive any vascular endothelial growth factor (VEGFR) inhibitor or Immune checkpoint blockade.
7. 18-75 years of age (inclusive)
8. Body weight≥40Kg
9. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
10. Patients capable of taking oral medication
11. Patients with evaluable or measurable lesions as per RECIST version 1.1
12. Expected survival >12 weeks

Exclusion Criteria:

1. with MSI-H colorectal adenocarcinoma as defined per local assessment using standard of care testing
2. Previous treatment with Fruquintinib or immune checkpoint inhibitors
3. Absolute neutrophil count (ANC)<1.5×109/L, or blood platelet count (PLT)<100×109/L, or hemoglobin<90g/L; blood transfusion within 1 week before enrollment for the purpose of enrollment is not allowed;
4. Serum total bilirubin>1.5×Upper Limit of Normal (ULN);Alanine transaminase(ALT) and/or Aspartate transferase (AST)>2.5×ULN (subject to the normal value at each site); or ALT and/or AST > 5×ULN for patients with liver metastases;
5. Creatinineclearancerate< 50mL/min;
6. Uncontrolled hypertension by monotherapy, i.e. systolic blood pressure >140mmHg or diastolic blood pressure >90mmHg after monotherapy treatment.
7. Clinical significant electrolyte abnormality;
8. Results of urine protein detection with 2+ or above, or urinary protein quantity ≥1.0g/24h;
9. Unrecovered toxicity fromprevious anticancer therapies(NCI CTC AE>Grade 1, except for alopecia and ≤Grade 2 neurotoxicity caused by Oxaliplatin), not fully recovered from previous surgeries; or the time from the last anticancer therapy or surgery is less than 4 weeks;
10. Central Nervous System (CNS) metastatic disease or prior cerebral metastasis;
11. Subjects with presence of clinically detectable second primary malignant tumors at enrollment, or other malignant tumors within the last 5 years (excluding adequately treated skin basal cell carcinoma or carcinoma in situ of cervix).
12. Clinically uncontrolled active infection, such as acute pneumonia, active hepatitis B or hepatitis C(previous medical history of hepatitis B virus infection regardless of drug control, HBV DNA≥104×copynumberor ≥2000IU/mL);
13. Difficulty in swallowing or known drug malabsorption;
14. Duodenal ulcer, ulcerative colitis, intestinal obstruction, other gastrointestinal diseases or other conditions that may lead to gastrointestinal bleeding or perforation according to the investigator's judgment; or with a history of intestinal perforation or intestinal fistula, which were not fully recovered after surgery;
15. History of artery thrombosis or deep venous thrombosis within 6 months before enrollment, or have evidence or a history of bleeding tendency within 2 months before the enrollment, regardless of severity;
16. Occurrence of stroke or transient ischemic attack within 12 months before the enrollment;
17. Activated Partial Thromboplastin Time (APTT) and/or prothrombin time (PT) > 1.5×ULN (subject to the normal range at each site);
18. Skin wounds, surgical site, trauma site, severe mucosal ulcers or fracture not completely healed;
19. Acute myocardial infarction, severe/unstable angina or received coronary artery bypass surgery within 6 months prior to enrollment; or patients with cardiac insufficiency of NYHA Grade 2 or above;
20. Pregnant or lactating women Or female subjects with childbearing potentials with positive pregnancy test result before the first time of study drug treatment;
21. Any clinical or laboratory abnormalities or compliance concerns unfit to participate in this clinical trial according to the investigator's judgment;
22. Serious psychological or psychiatric disorders;
23. Contraindications of immune checkpoint inhibitors
24. Participated in any other drug clinical trial during the last 4 weeks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
PFS(progression free survival) rate at 6 months | 6 months
  To determine the clinical effectiveness of the study treatment assessed using PFS rate at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China